CLINICAL TRIAL: NCT02688712
Title: Phase II Study of TGFβ Type I Receptor Inhibitor LY2157299 With Neoadjuvant Chemoradiation in Patients With Locally Advanced Rectal Adenocarcinoma
Brief Title: ExIST Study of LY2157299 (Galunisertib) in Rectal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-050A
Record Dates: First submitted 2016-01-25; First posted 2016-02-23 (Estimated); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Rectal Adenocarcinoma
Keywords: IIA; Xeloda; radiation therapy; LY2157299; tumor resection; capecitabine; 5FU; Fluorouracil; IIB; IIC; IV; neoadjuvant; Rectal cancer; Immunotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — LY-2157299; Capecitabine; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2157299 + Chemoradiation + Surgery (Experimental): Patients will receive a 14 day course of LY2157299. On day 15 patients will begin chemoradiation treatment with Capecitabine or Fluorouracil. On day 29, patients will undergo another fourteen day course of LY2157299 concurrent with their ongoing chemoradiation treatment. Six to ten weeks after completing their neoadjuvant therapy, patient will undergo a tumor specific mesorectal excision as per standard of care.
  Interventions: Drug: LY2157299; Drug: Capecitabine; Drug: Fluorouracil; Procedure: Tumor specific mesorectal excision

INTERVENTIONS:
Drug: LY2157299 — Small molecule inhibitor of transforming growth factor-beta signaling pathway
  Other Names: Galunisertib
Drug: Capecitabine — Antimetabolite chemotherapy
  Other Names: Xeloda
Drug: Fluorouracil — Antimetabolite chemotherapy
  Other Names: 5-fluorouracil , 5-FU, Adrucil, Efudex, Fluoroplex
Procedure: Tumor specific mesorectal excision — Tumor specific mesorectal excision

SUMMARY:
The purpose of this study is to see how effective and safe LY2157299, in combination with chemotherapy and radiation therapy, might be in treating rectal cancer. Also as part of this study, research will be done on tumor samples to see if it is possible to predict if patients will respond to treatment, and blood samples to look at the immune system response to study treatment.

About 50 people will take part in this study. The study treatment will be given over an 8 week period and the investigators will continue to collect your health information for up to 5 years, as part of this study

DETAILED DESCRIPTION:
This is a prospective Phase II study to test the efficacy of LY2157299 in combination with neoadjuvant chemoradiation in patients with rectal adenocarcinoma. This study will test the hypothesis that LY2157299 will improve effector T cell tumor infiltration and activity resulting in improved pathologic response rates. The investigators propose that this improved immune response will result in improved disease-free and overall survival.

The objectives are:

1. Determine the rate of pathologic complete response in patients with locally advanced rectal adenocarcinoma treated with neoadjuvant chemoradiation and the investigational agent LY2157299
2. Correlate immunoscore changes prior to therapy, during therapy, and at surgical resection with pathologic response and MRI parameters
3. Immune monitoring to evaluate potential biomarkers of treatment success.

Eligible patients will have histologically confirmed rectal adenocarcinoma, AJCC Stage IIA IIIC or AJCC Stage IV appropriate for consideration of primary rectal tumor resection. Patients will undergo a forceps biopsy of the rectal mass as part of the diagnostic workup as well as undergo staging evaluation including an MRI with additional study sequences. Enrolled patients will receive a 14 day course of LY2157299 followed by a repeat biopsy and MRI with study sequences. In this trial the investigators plan to use the maximum tolerated dose of LY2157299 established in human clinical trials, 300mg delivered as 150mg P.O. BID. On day 15 patients will begin chemoradiation with either 5-FU (fluorouracil ) or capecitabine (Xeloda®). On day 29, patients will undergo another fourteen day course of LY2157299 concurrent with their ongoing chemoradiation.

Patients will undergo 50.4 to 54Gy of radiation in 1.8Gy daily fractions delivered Monday through Friday for a total of 28-30 fractions. The acceptable duration of chemoradiation, including treatment breaks or delays, is up to 8 weeks total. Six to ten weeks after completing their neoadjuvant therapy, patient will undergo a tumor specific mesorectal excision as per standard of care with evaluation of pathologic response rate. Patients will be followed for disease-free survival, progression free survival, local recurrence, and overall survival. A three patient safety lead-in will be performed, where a six week safety period following completion of radiation will be completed prior to enrolling subsequent patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients (male and female) with histologically confirmed rectal adenocarcinoma, AJCC Stage IIA-IIIC or AJCC Stage IV appropriate for consideration of primary rectal tumor resection.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Age 18 years or above.
* Laboratory values (performed within 28 days prior to enrollment) as follows:

  * WBC ≥3.0 109/L
  * Hgb ≥9g/dl (patients may be transfused to reach this level)
  * Platelets ≥99 109 /L
  * Creatinine ≤1.5X upper limit of laboratory normal
  * AST/ALT ≤5 X upper limit of laboratory normal
  * Total bilirubin ≤1.5X upper limit of laboratory normal
  * BNP ≤ 3 times the baseline value and upper limit of laboratory normal
  * Troponin I ≤ upper limit of laboratory normal
  * hsCRP ≤ upper limit of laboratory normal
  * Cystatin ≤ upper limit of laboratory normal
  * PT/INR ≤1.5X upper limit of laboratory normal
* Pre-menopausal women must have a negative pregnancy test on the day treatment starts and must avoid becoming pregnant while on treatment and for 3 months following completion of therapy. Men must avoid fathering a child while on treatment and for 3 months following completion of therapy. This exclusion is required due to the toxicities that chemotherapy, radiation, and LY2157299 may have on the forming fetus, spermatogenesis or the nursing child. Also, because pregnancy may alter immune function it may limit the treatment efficacy. Women of childbearing potential must agree to use a medically approved contraceptive method during the treatment period and for 3 months following the last dose of LY2157299. Contraceptive methods may include an intrauterine device [IUD], birth control pills or barrier method. If condoms are used as a barrier method, a spermicidal agent should be added as a double barrier protection.
* No active bleeding.
* Ability to give informed consent and comply with the protocol. Patients with a history of psychiatric illness must be judged able to understand fully the investigational nature of the study and the risks associated with the therapy.

Exclusion Criteria:

* Active infection requiring systemic antibiotics.
* Active autoimmune disease as defined by the autoimmune disease assessment tool (see protocol)
* Diagnosis of a solid tumor malignancy (excluding non-melanoma skin cancer) within 3 years of enrollment.
* History of prior pelvic radiation.
* Aortic aneurysm (see protocol)
* Abnormal Echocardiogram (see protocol)
* Immunodeficiency, need for immunosuppressive medications, or need for chronic steroids.
* Participation in any investigational drug study within 28 days of enrollment.
* Pregnant or lactating women, as treatment involves risks to the embryo or fetus.
* Other medical or psychiatric conditions that in the opinion of the Principal Investigator would preclude safe participation in protocol.
* History of cardiac disease, including myocardial infarction within 6 months before study entry, unstable angina pectoris, New York Heart Association Class III/IV congestive heart failure, or uncontrolled hypertension, major cardiac abnormalities, a predisposition for developing aneurysms including family history of aneurysms, Marfan syndrome, bicuspid aortic valve, or evidence of damage to the large vessels of the heart.
* Concomitant use of strong CYP3A4 inhibitors and inducers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-03-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of pathologic response | Patients should be evaluated for response at surgery and every 3 months for 2 years and then every 6 months at year three and four. All patients will be followed for survival until death or 5 years post-treatment (whichever comes first)
  Complete response is defined as no viable tumor cells identified.

SECONDARY OUTCOMES:
Immunoscore (utilizing tumor tissue) | Screening Visit, Day 15 Visit and Day of Surgery
  For the immunoscore, a value of 0 or 1 is assigned to each cell population of interest with 0 corresponding to a poor immune infiltrate and 1 corresponding to a favorable immune infiltrate as determined by immunohistochemistry.
MRI Parameters | Screening Visit and Day 15 Visit
  Investigators will test a minimum of three MRI parameters including but not limited to ADC and f_p from the IVIM sequence, and Ktrans from the DCE sequence.
Immunologic monitoring parameters | Days 1, 15, 22, 29, 43, 57 Visits, and Day of Surgery.
  The immunologic monitoring parameters will be combined to arrive at an aggregated measure of "pro-tumor immune environment" or "anti-tumor immune environment" using cell counts derived from flow cytometry of peripheral blood and serum measures of inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Young, MD, PhD, Principal Investigator — Providence Health & Services; Todd Crocenzi, MD, Principal Investigator — Providence Health & Services
Locations (1):
- Providence Cancer Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yamazaki T, Gunderson AJ, Gilchrist M, Whiteford M, Kiely MX, Hayman A, O'Brien D, Ahmad R, Manchio JV, Fox N, McCarty K, Phillips M, Brosnan E, Vaccaro G, Li R, Simon M, Bernstein E, McCormick M, Yamasaki L, Wu Y, Drokin A, Carnahan T, To Y, Redmond WL, Lee B, Louie J, Hansen E, Solhjem MC, Cramer J, Urba WJ, Gough MJ, Crittenden MR, Young KH. Galunisertib plus neoadjuvant chemoradiotherapy in patients with locally advanced rectal cancer: a single-arm, phase 2 trial. Lancet Oncol. 2022 Sep;23(9):1189-1200. doi: 10.1016/S1470-2045(22)00446-6. Epub 2022 Aug 8. PMID 35952709
- See also: Providence Cancer Center Clinical Trials — http://oregon.providence.org/our-services/p/providence-cancer-center-clinical-trials/